CLINICAL TRIAL: NCT03459131
Title: Clinical Evaluation of Two Monthly Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLD523-E001
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BIOFINITY ENERGYS then BIOFINITY (Other): Comfilcon A with Digital Zone Optics™ contact lenses worn first, followed by comfilcon A contact lenses. Each product will be worn bilaterally (in both eyes) for 7 days in a daily wear modality.
  Interventions: Device: Comfilcon A with Digital Zone Optics™ contact lenses; Device: Comfilcon A contact lenses
- BIOFINITY then BIOFINITY ENERGYS (Other): Comfilcon A contact lenses worn first, followed by comfilcon A with Digital Zone Optics™ contact lenses. Each product will be worn bilaterally (in both eyes) for 7 days in a daily wear modality.
  Interventions: Device: Comfilcon A with Digital Zone Optics™ contact lenses; Device: Comfilcon A contact lenses

INTERVENTIONS:
Device: Comfilcon A with Digital Zone Optics™ contact lenses — Silicone hydrogel spherical contact lenses with Digital Zone Optics™
  Other Names: BIOFINITY® ENERGYS™
Device: Comfilcon A contact lenses — Silicone hydrogel spherical contact lenses
  Other Names: BIOFINITY®

SUMMARY:
The purpose of this study is to explore overall vision with BIOFINITY® ENERGYS™ contact lenses as compared to BIOFINITY® contact lenses after one week of wear.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an approved informed consent form (ICF);
* Successful wear of BIOFINITY® (spherical) (or private label) contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months;
* Best-corrected visual acuity (BCVA) 20/25 or better in each eye;
* Possess spectacles that provide a corrected visual acuity of 20/40 or better in both eyes (OU) and be willing to wear them (as needed);
* Currently using digital devices (computer, tablet, and/or smart phone) for a minimum of 5 days per week and 4 hours per day;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any anterior segment infection, inflammation, abnormality or disease that contraindicates contact lens wear;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated;
* Refractive, ocular, or intraocular surgery, as specified in the protocol;
* Current or history of eye injury or disorders, as specified in the protocol;
* Current or history of intolerance, hypersensitivity or allergy to any component of the study products;
* Habitual contact lens wear in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment;
* Use of topical ocular medications that would require instillation during contact lens wear;
* Other protocol-specified exclusion criteria may apply.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, A Novartis Division, Study Director — Alcon, A Novartis Division
Locations (1):
- Alcon Investigative Site, Maitland, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from one study site located in the US.
Pre-assignment Details: All 15 enrolled subjects were randomized and exposed to investigational product. This reporting group includes all randomized and treated subjects (15).
Period: Period 1, First 7 Days of Wear
Arm/Group | BIOFINITY ENERGYS Then BIOFINITY | BIOFINITY Then BIOFINITY ENERGYS
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Period 2, Second 7 Days of Wear
Arm/Group | BIOFINITY ENERGYS Then BIOFINITY | BIOFINITY Then BIOFINITY ENERGYS
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study (Safety Analysis Set).
Groups:
- Overall: Comfilcon A with Digital Zone Optics™ contact lenses and comfilcon A contact lenses worn during Period 1 and Period 2 in a crossover assignment, as randomized.
Arm/Group | Overall
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14
  Black or African American | 0
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 1
  Multi-Racial | 0

OUTCOME MEASURES:

1. Primary Outcome: Subjective Rating of Overall Vision
Description: Overall vision was assessed binocularly (both eyes together) by the subject on a 10-point scale, where 1=poor and 10=excellent. Inferential testing was not planned for this primary effectiveness endpoint.
Time Frame: Day 7, each product
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- BIOFINITY ENERGYS: Comfilcon A with Digital Zone Optics™ contact lenses worn during Period 1 or Period 2 for 7 days.
- BIOFINITY: Comfilcon A contact lenses worn during Period 1 or Period 2 for 7 days.
Arm/Group | BIOFINITY ENERGYS | BIOFINITY
Number analyzed (Participants) | 15 | 15
units on a scale | 8.6 (1.2) | 8.6 (1.1)

2. Secondary Outcome: Over-refraction
Description: Over-refraction (amount of additional correction needed to improve visual acuity (VA)) was collected for each eye and measured in diopters (D). Inferential testing was not planned for this endpoint.
Time Frame: Day 1 (Dispense), each product
Population: Safety Analysis Set
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | BIOFINITY ENERGYS | BIOFINITY
Number analyzed (Participants) | 15 | 15
Number analyzed (Eyes) | 30 | 30
Eyes
  -0.25D | 3 | 0
  0.00D | 26 | 24
  +0.25D | 1 | 6

ADVERSE EVENTS:
Time Frame: Dispense through study completion, an average of 14 days
Description: An Adverse Event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device. Safety Analysis Set, based on treatment-specific exposure. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.
Groups:
- BIOFINITY ENERGYS: All subjects exposed to comfilcon A with Digital Zone Optics™ contact lenses
- BIOFINITY: All subject exposed to comfilcon A contact lenses
Arm/Group | BIOFINITY ENERGYS | BIOFINITY
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03459131/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03459131/SAP_001.pdf